CLINICAL TRIAL: NCT00352612
Title: Comparison of Cephalexin Versus Clindamycin in the Empiric, Outpatient Treatment of Suspected Staphylococcal Cutaneous Infections in the Era of Community-associated Methicillin-resistant Staphylococcus Aureus (CA-MRSA)
Brief Title: Comparison of Cephalexin Versus Clindamycin for Suspected CA-MRSA Skin Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aaron Chen (Other)
Collaborators: Thrasher Research Fund (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Aaron Chen, MD, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00003301
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-04

CONDITIONS: Staphylococcal Infection; Abscess; Staphylococcal Skin Infection; Folliculitis
Keywords: clinical trial; randomized; blinded; controlled
MeSH Terms: conditions — Staphylococcal Infections; Abscess; Staphylococcal Skin Infections; Folliculitis | interventions — Clindamycin; Cephalexin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cephalexin (Placebo Comparator)
  Interventions: Drug: cephalexin
- clindamycin (Active Comparator)
  Interventions: Drug: clindamycin

INTERVENTIONS:
Drug: clindamycin — clindamycin suspension or tablets, 20mg/kg/day, given by mouth, divided TID, for 7 days
  Arms: clindamycin
Drug: cephalexin — cephalexin suspension or tablets, 40mg/kg/day, given by mouth, divided TID, for 7 days
  Other Names: keflex
  Arms: cephalexin

SUMMARY:
The purpose of this study is to help define the role of antibiotics in the treatment of pediatric skin infections caused by community-associated methicillin-resistant Staphylococcus aureus (CA-MRSA). The investigators hypothesize that treatment with cephalexin, a penicillin-like antibiotic to which CA-MRSA would be expected to be resistant, does not result in poorer outcomes than treatment with clindamycin, an antibiotic to which CA-MRSA is most often susceptible.

DETAILED DESCRIPTION:
Community-associated methicillin resistant Staphylococcus Aureus (CA-MRSA) infections have increased significantly over the past decade. Nearly every major region of the country has reported infections with this organism, with some areas reporting a prevalence as high as 80%. Epidemiologic evidence points to the emergence of a new strain of MRSA within the community, with unique genetic and clinical characteristics that differentiate it from traditional hospital-associated MRSA (HA-MRSA). Unlike HA-MRSA, these CA-MRSA are often susceptible in vitro to multiple antibiotic classes (other than penicillins and cephalosporins), and often cause significant, deep-seated abscesses in healthy individuals without any known risk factors for healthcare contact. Prior to awareness of this disease, many clinicians were using penicillin and cephalosporin antibiotics for empiric treatment of cutaneous abscesses, yet widespread treatment failures in the face of increasing CA-MRSA infections did NOT occur. During a one-year retrospective study in pediatric patients at our institution, we found that nearly 50% of CA-MRSA abscesses were treated with "inappropriate" antibiotics by susceptibility profiles without any significant adverse outcomes. Many clinicians are now confronted with the dilemma of whether to change empiric antibiotic therapy to other classes to which CA-MRSA would be expected to be susceptible; the most common choices including clindamycin, trimethoprim-sulfamethoxazole (TMP-SMX), or vancomycin. Unfortunately, each of these antibiotics has problems of its own in terms of increased cost, poor palatability of pediatric liquid formulation, poorer side effect profile, or necessity of IV infusion, and at this time the optimal, empiric antibiotic treatment for presumed CA-MRSA skin and soft tissue infections is unclear.

The purpose of this study is to help define the role of antibiotics in the treatment of pediatric skin infections caused by CA-MRSA. We hypothesize that treatment with cephalexin, a penicillin-like antibiotic to which CA-MRSA would be expected to be resistant, does not result in poorer outcomes than treatment with clindamycin, an antibiotic to which CA-MRSA is most often susceptible.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 months and 18 years of age (inclusive)
* Suspected purulent staphylococcal skin or soft tissue infection
* No hospitalization within the previous 14 days
* Must have reliable means of follow-up contact (e.g. working phone)
* Outpatient management in the judgement of treating physician

Exclusion Criteria:

* Hospitalization on initial visit
* Voluntary withdrawal by the treating physician in order to dictate the antibiotic being used
* Patients with a history of hypersensitivity to or intolerance of cephalexin (or other beta lactams) or clindamycin.
* Patients with altered immunity (inherited or acquired)
* Patients with skin infections related to surgical wounds or hardware.
* Patients currently on antibiotic therapy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Chen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cephalexin: patients who received cephalexin
- Clindamycin: those who received clindamycin
Period: Overall Study
Arm/Group | Cephalexin | Clindamycin
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: cephalexin arm
- Group 2: clindamycin arm
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 100 | 200
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 60 | 115
  Male | 45 | 40 | 85

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement at the 48-72 Hour Clinical Follow-up
Description: Clinical improvement was defined as improvement in at least one of the following four measures without regression in any: (1) erythema (2) pain (3) induration (4) patient or families self report of improvement.
Time Frame: 48-72 hour clinical follow-up
Measure: Number; unit: participants
Groups:
- Cephalexin: those patients who received cephalexin
- Clindamycin: those patients who received clindamycin
Arm/Group | Cephalexin | Clindamycin
Number analyzed (Participants) | 100 | 100
participants | 94 | 97

ADVERSE EVENTS:
Arm/Group | Cephalexin | Clindamycin
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes